CLINICAL TRIAL: NCT05781971
Title: Department of Intensive Care Medicine, The First Affiliated Hospital of Soochow University
Brief Title: Effect of Nutritional Support and Early Rehabilitation on Sepsis
Acronym: NUSPOTER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Yao Wei,MD, associate chief physician, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NUSPOTER
Record Dates: First submitted 2023-02-01; First posted 2023-03-23 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Life Quality; Hospital Mortality
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- high protein + early bedside rehabilitation (Experimental)
  Interventions: Dietary Supplement: high protein; Behavioral: rehabilitation
- high protein alone (Active Comparator)
  Interventions: Dietary Supplement: high protein
- standard protein + early bedside (Placebo Comparator): standard protein and rehabilitation
  Interventions: Behavioral: rehabilitation; Dietary Supplement: standard protein
- standard protein (Sham Comparator): only standard protein
  Interventions: Dietary Supplement: standard protein

INTERVENTIONS:
Dietary Supplement: high protein — Patients in high-protein group will be given a target protein amount of 2.0 g/kg/d. Standard enteral nutrition is the first choice,the remaining target value will be met by intravenous amino acid infusion.
  Arms: high protein + early bedside rehabilitation; high protein alone
Behavioral: rehabilitation — In this trial, the investigator will provide early rehabilitation treatment such as respiratory training, bicycle training, and medium frequency electrical stimulation to patients.
  Arms: high protein + early bedside rehabilitation; standard protein + early bedside
Dietary Supplement: standard protein — The investigator set a protein target of 1.2 g/Kg/d for the standard protein group, which will be supplied enterally or parenterally.
  Arms: standard protein; standard protein + early bedside

SUMMARY:
Sepsis is a syndrome of life-threatening organ dysfunction caused by a dysregulated host response to infection.Acute catabolic response in critically ill patients struck by sepsis, manifested by massive protein breakdown in a short time.This pathology frequently leads to prolonged hospitalization and mechanical ventilation, increased mortality, and reduced quality of survival.It is uncertainty whether sepsis patients in ICU can benefit from high protein intake combined with early exercise. Even though the combination has been shown to be beneficial in other populations.In the present study, the investigator will evaluate the effects of a combination of high protein targets combined with early rehabilitation in sepsis patients in ICU.

DETAILED DESCRIPTION:
Existing research results confirm that high target protein support can reduce the mortality of sepsis patients. Early bedside rehabilitation has a good effect on cognitive function after ICU. This study combined high-protein nutritional support with bedside rehabilitation to improve the quality of life in patients with sepsis after ICU.

ELIGIBILITY:
Inclusion Standard

1. Patients with sepsis
2. Patients aged 18-70 years
3. Time of admission ≤48 h
4. Non-terminal condition

Exclusion Standard

1. Severe acute kidney injury
2. Severe chronic liver disease (MELD score ≥20) or acute hepatic failure
3. Protein allergy
4. Pregnancy and lactation
5. BMI≥30 kg/m²

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Hospital Mortality | Day 90
  Chart review

SECONDARY OUTCOMES:
Nutrition related indicators | Hospital discharge
  Chart review
Physical functioning | Hospital discharge
  Grip dynamometer
Prognostic factor | Hospital discharge
  Chart review
Health-related quality of life | Day 90
  SF-36 and EQ-5D-5L

IPD SHARING:
Plan to Share IPD: Undecided